CLINICAL TRIAL: NCT01891799
Title: Situkulwane Lesiphephile-Safe Generations: Improving Approaches to Antiretroviral Therapy for HIV-Positive Pregnant Women
Brief Title: Swaziland Safe Generations
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Ministry of Health, Swaziland (Other Government); University of Cape Town (Other); Elizabeth Glaser Pediatric AIDS Foundation (Other); National Emergency Response Council on HIV and AIDS (NERCHA) (Unknown)
Responsible Party: Principal Investigator, Elaine J. Abrams, MD, Professor of Epidemiology, Columbia University
Other Study IDs: AAAL0661; AID-OAA-A-12-000020 (Other Grant/Funding Number: USAID)
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; PMTCT; Option B+; Swaziland
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — 50 microliters of capillary blood will be drawn via heelstick or finger prick phlebotomy from infants using filter paper. Blood will be collected from infants at 6mos of age to conduct DNA PCR HIV testing, specifically for this study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PMTCT Options Evaluation: All HIV positive pregnant women not on ART engaging in PMTCT services at the study sites will be included. This will include HIV+ women not on ART enrolling in PMTCT services and pregnant women newly testing HIV+ in the ANC. All women will eventually receive the intervention of Option B+ as each clinic transitions from Option A to B+.
  Interventions: Other: Option B+

INTERVENTIONS:
Other: Option B+ — * Using one low toxicity triple ARV regimen [(tenofovir (TDF) + lamivudine/emtricitabine (3TC/FTC) + efavirenz (EFV)] for all women, rather than adapting regimens by CD4+
  * Engaging all pregnant and postpartum women and their infants in the structured appointment and follow-up system currently only available to women receiving ART
  * Providing a simplified standardized public health approach both antenatally and postnatally, with adherence and retention support tailored to the particular health and social needs of peripartum women

SUMMARY:
The purpose of this study is to understand how best to provide care and treatment services to human immunodeficiency virus (HIV) positive pregnant women and their babies in Swaziland. The study is designed to evaluate a new approach for Preventing Mother-to-Child Transmission (PMTCT)where all HIV positive pregnant women initiate lifelong triple antiretroviral (ARV) therapy regardless of their disease stage. The goal is to prevent delays in women accessing treatment for their own health and ensure that women and their children remain in care. This study will compare this new approach to PMTCT, known as Option B+, to Option A, which is the current standard of care for PMTCT in Swaziland. The study will be conducted at 10 health facilities in the Manzini and Lubombo regions in Swaziland. The study has three components: the main component is a PMTCT Options Evaluation where data from medical records will be abstracted on all HIV positive pregnant women attending antenatal services at the 10 selected study facilities; data will be abstracted on their HIV exposed infants as well. Other components of the study include a PMTCT Options Acceptability Evaluation using semi-structured questionnaires with PMTCT clients and health care workers (HCWs) as well as a cost effectiveness evaluation comparing costs under conditions of Option A and Option B+.

DETAILED DESCRIPTION:
Purpose:

"Situkulwane Lesiphephile-Safe Generations" is an implementation science research study designed to evaluate an innovative PMTCT strategy that includes a modified Option B approach, where all HIV positive pregnant women initiate lifelong triple antiretroviral (ARV) therapy independent of CD4+ count (Option B+) and all HIV positive pregnant and postpartum women and their infants are engaged in the same structured appointment and follow-up protocols currently available only to women receiving antiretroviral therapy (ART). The study hypothesizes that this single, uniform and streamlined treatment and retention approach for all HIV positive pregnant women will eliminate delays, prevent losses and will: (1) result in a higher proportion of mothers and infants successfully completing the PMTCT cascade and fewer new pediatric infections; (2) lead to a higher proportion of ART-eligible women initiating triple ART earlier in pregnancy; (3) will be more feasible to implement; 4) have greater acceptability among staff and patients; and 5) will be more cost-effective compared to Option A.

Design:

Stepped wedge design at 10 health facilities with one facility transitioning from Option A to the Option B+ approach every month over 12 months. Outcome measures will be compared under Option A and Option B+ conditions for all sites as well as before and after the transition at each site. Routinely collected data from facility registers and medical records will be abstracted to determine study outcomes. In addition, two purposely selected cohorts of (1)120 PMTCT clients and; (2) approximately 50 health care workers will complete questionnaires at repeated time points to assess acceptability of Option A and Option B+ approaches.

Study Population:

All HIV positive pregnant women not on ART engaging in PMTCT services at the study sites will be part of the PMTCT Options Evaluation. This will include HIV+ women not on ART enrolling in PMTCT services and pregnant women newly testing HIV+ in the absolute neutrophil count (ANC). A subset of HIV+ pregnant women not on ART engaging in PMTCT services and health care workers providing PMTCT services at the study sites will be enrolled in an acceptability evaluation.

Study Size:

A total of approximately 2,600 HIV positive pregnant women enrolled in PMTCT services at ten Ministry of Health (MOH) facilities.

Primary Objective:

To compare the impact of implementing Option A and Option B+ on the composite endpoint of infant HIV-positive polymerase chain reaction (PCR) at 6 months postpartum or maternal loss to follow-up at 6 months postpartum.

Secondary Objectives:

1. To compare Option A and Option B+ on proportion of pregnant women with CD4+<350 cells/mm3 initiating ART during pregnancy and on duration of ART received prior to delivery for ART-eligible pregnant women
2. To compare Option A and Option B+ on the proportion of women and children retained in HIV care at 12, and 18 months postpartum
3. To examine patient and provider level acceptability of Option A and Option B+
4. To compare the cost-effectiveness of Option A and Option B+

Tertiary Objectives:

1. To determine pregnancy and infant outcomes (including fetal losses, neonatal death, birth weight and gestational age) among HIV+ pregnant women receiving PMTCT and compare outcomes by maternal ARV regimens.
2. To compare Option A and Option B+ on maternal and child adherence as measured by prescriptions dispensed for maternal and infant antiretroviral medications.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 18 years of age
* Documented pregnancy (per routine ANC protocol in this setting)
* Documented HIV-infection (per routine ANC protocol in this setting)
* Infants born to eligible and enrolled women

Exclusion Criteria:

• Women already on ART when entering ANC

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for the PMTCT Options Evaluation is all HIV+ pregnant women not on ART at their first ANC visit at the 10 study facilities. A total of approximately 2600 mother-infant pairs (2600 HIV positive women + 2600 of their HIV exposed babies) will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 2518 (Actual)
Dates: Start 2013-08; Primary Completion 2016-10-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Number of (1) infant HIV positive PCR at six months postpartum OR (2) mother lost to follow-up from at six months postpartum | Up to 24 months
  Combined maternal-child endpoint: The primary outcome will be measured on all HIV+ pregnant women not on ART at their first ANC visit at a participating study site, approximately 2600 women(becoming mother-infant pairs postpartum). This includes women entering PMTCT with known HIV+ status, not on ART, and women testing HIV+ on entry into ANC.

SECONDARY OUTCOMES:
Proportion of pregnant women with CD4+<350 cells/mm3 initiating ART during pregnancy | Up to 24 months
  ART Initiation During Pregnancy: Proportion of pregnant women with CD4+<350 cells/mm3 initiating ART during pregnancy
Proportion of women and children retained in HIV care at 12 and 18 months postpartum | Up to 24 months
  Maternal/Infant Retention in Care: Proportion of women and children retained in HIV care at 12 and 18 months postpartum
Duration of ART/ARV received prior to delivery | Up to 24 months
  ART/ARV Duration: Duration of ART/ARV received prior to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Elaine J Abrams, MD, Principal Investigator — Columbia University
Locations (12):
- Eswatini (12):
  - Good Shepherd Hospital, Siteki, Lubombo Region
  - Siphofaneni, Siteki, Lubombo Region
  - Siteki PHU, Siteki, Lubombo Region
  - Family Life Association Clinic, Manzini
  - King Soghuza II PHU, Manzini
  - Lamvelase Clinic, Manzini
  - Luyengo Clinic, Manzini
  - Mankayane PHU, Manzini
  - Mbabane Government Hospital, Manzini
  - Mbikhwakhe Clinic, Manzini
  - MSF Matsapha, Manzini
  - Raleigh Fitkin Memorial Hospital, Manzini

REFERENCES:
- [Derived] DiCarlo AL, Gachuhi AB, Mthethwa-Hleta S, Shongwe S, Hlophe T, Peters ZJ, Zerbe A, Myer L, Langwenya N, Okello V, Sahabo R, Nuwagaba-Biribonwoha H, Abrams EJ. Healthcare worker experiences with Option B+ for prevention of mother-to-child HIV transmission in eSwatini: findings from a two-year follow-up study. BMC Health Serv Res. 2019 Apr 2;19(1):210. doi: 10.1186/s12913-019-3997-1. PMID 30940149